CLINICAL TRIAL: NCT01045135
Title: The Effect of Pregnancy and Labour on the Pelvic Floor Diagnosed With 3D and 4D Ultrasound
Status: Completed | Type: Observational
Sponsor: University Hospital, Akershus (Other)
Collaborators: The Research Council of Norway (Other); South-Eastern Norway Regional Health Authority (Other)
Responsible Party: Principal Investigator, Marie Ellstrøm Engh, M.D. PhD, University Hospital, Akershus
Other Study IDs: Pelvic floor ultrasound
Record Dates: First submitted 2010-01-07; First posted 2010-01-08 (Estimated); Results first posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Obstetric; Injury Pelvic Floor
Keywords: Pelvic organ prolapse; Levator hiatus; 3 and 4 dimensional ultrasound
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- first time delivery: Women giving birth to their first child

SUMMARY:
Injuries to the pelvic floor muscles and fascias during delivery and childbirth may lead to urinary incontinence (25-45 %), faecal incontinence (11-45%), pelvic organ prolapse (7-23%), sexual dysfunction (15-33 %) and chronic pain syndromes (4-15%). Pelvic floor muscle injuries are not easy to diagnose as they are not visible when looking at surface anatomy during a standard gynaecological examination. The investigators are therefore in urgent need of better tools to diagnose these injuries. Having a reliable and easily accessible tool enables studies of the consequences of such pelvic floor muscle injuries. It also makes it possible for us to explore the effect of interventions such as pelvic floor muscle training and surgery in patients with and without pelvic floor muscle injuries. The investigators have previously presented data to support the reliability and the validity of the three and four dimensional (3 and 4D) ultrasound technique used to define pelvic floor muscle anatomy in healthy volunteers and have now a tool to study women before and after delivery. At the Department of Obstetrics and Gynaecology, Akershus University Hospital there are approximately 4500 deliveries annually and 1500 women are giving birth for the first time.

Challenges: The invitation to participate in the study will be given to all women expecting their first child fulfilling inclusion criteria. The biggest challenges in the project will be logistical. To be able to inform, recruit and follow women having their first child is a challenge in it self.

Applications: If it is possible to identify a risk group for pelvic floor injuries before delivery, it might be ethical to recommend a prophylactic caesarean section to avoid disabling incontinence and prolapse later in life.

ELIGIBILITY:
Inclusion Criteria:

* Women giving birth to their first child at Akershus University Hospital, Norway
* Must understand spoken and written Norwegian

Exclusion Criteria:

* Previous pregnancy of more than 16 weeks
* Serious illness mother or child
* Birth before pregnancy week 32

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women giving birth to their first child at Akershus University Hospital, Norway
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2009-12; Primary Completion 2012-10 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie E Engh, M.D., PhD, Study Director — University Hospital, Akershus
Locations (1):
- Akershus University Hospital, Lørenskog, Akershus, Norway

REFERENCES:
- [Derived] Bo K, Hilde G, Staer-Jensen J, Siafarikas F, Tennfjord MK, Engh ME. Does general exercise training before and during pregnancy influence the pelvic floor "opening" and delivery outcome? A 3D/4D ultrasound study following nulliparous pregnant women from mid-pregnancy to childbirth. Br J Sports Med. 2015 Feb;49(3):196-9. doi: 10.1136/bjsports-2014-093548. Epub 2014 Aug 6. PMID 25100734

RESULTS

PARTICIPANT FLOW:
Recruitment Details: January 2010 - july 2011
Period: Overall Study
Arm/Group | First Time Delivery
Started | 300
Completed | 274
Not Completed | 26

BASELINE CHARACTERISTICS:
Arm/Group | First Time Delivery
Number analyzed (Participants) | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 300
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.6 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 300
  Male | 0
Region of Enrollment [Number; unit: participants]
  Norway | 300

OUTCOME MEASURES:

1. Primary Outcome: Change in Levator Hiatus Area at Rest Measured Via 3-dimensional Ultrasound at Gestational Week 21 and 37.
Description: 3-dimensional ultrasound was used to capture the axial plane of the pelvic floor in order to measure LH area. Levator hiatus area was measured at gestational week 21 and 37, at rest, during contraction and during Valsalva maneuver - giving 6 measurements all together. The change in LH area was computed between the two different timepoints giving 3 outcomes
Time Frame: 21 weeks and 37 weeks of gestation
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Primiparous Women Levator Hiatus Area During Valsalva Maneuver: Women giving birth to their first child
Arm/Group | Primiparous Women Levator Hiatus Area During Valsalva Maneuver
Number analyzed (Participants) | 274
cm | 2.0 (1.7)

2. Primary Outcome: Change in Levator Hiatus Area at Contraction Measured Via 3D Ultrasound at Gestational Week 21 and 37
Description: 3-dimensional ultrasound was used to capture the axial plane of the pelvic floor in order to measure LH area. Levator hiatus area was measured at gestational week 21 and 37, at rest, during contraction and during Valsalva maneuver - giving 6 measurements all together. The change in LH area was computed between the two different timepoints.
Time Frame: 21 weeks and 37 weeks of gestation
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Primiparous Women Bladder Neck Mobility Rest to Valsalva Maneu: Women giving birth to their first child
Arm/Group | Primiparous Women Bladder Neck Mobility Rest to Valsalva Maneu
Number analyzed (Participants) | 274
cm | 1.2 (1.2)

3. Other Pre Specified Outcome: Health Related Complaints
Time Frame: 20 months
Reporting Status: Not Posted

4. Primary Outcome: Change in Levator Hiatus Area During Valsalva Maneuver Measured Via 3D Ultrasound
Description: as for outcome 2
Time Frame: gestational week 21 and 37
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Primiparous Women Levator Hiatus Area: Women giving birth to their first child
Arm/Group | Primiparous Women Levator Hiatus Area
Number analyzed (Participants) | 274
cm | 3.3 (3.5)

5. Secondary Outcome: Change in Bladder Neck Mobility Measured Via 3D Ultrasound
Description: 3-dimensional ultrasound was used to capture the axial plane of the pelvic floor in order to measure LH area. Bladder neck mobility was measured at gestational week 21 and 37, at rest and during Valsalva maneuver . The change in mobility from rest to valsalva was computed between the two different timepoints.
Time Frame: gestational week 21 and 37
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Primiparous Women Bladder Neck Mobility Rest to Valsalva Maneu
Number analyzed (Participants) | 274
cm | -0.11 (0.8)

ADVERSE EVENTS:
Description: Serious and other (non-serious) adverse effects were not collected/assessed, as this was an observational cohort study with no intervention.
Arm/Group | First Time Delivery
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
We did not examine the women before they were pregnant and therefore do not have information about how the pelvic floor was before pregnancy.

It is therefore possible that we have underestimated the change happening to the levator hiatus.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No